CLINICAL TRIAL: NCT05328843
Title: An Open-label Phase I Clinical Study to Evaluate the Pharmacokinetic Characteristics of Single-dose of Pegylated Exenatide Injection (PB-119) in Subjects With Different Degrees of Renal Insufficiency and Matched Subjects With Normal Renal Function
Brief Title: Study to Evaluate the Pharmacokinetic Characteristics of Pegylated Exenatide Injection (PB-119) in Subjects With Different Degrees of Renal Insufficiency and Matched Subjects With Normal Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB119109
Record Dates: First submitted 2022-04-05; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Type2Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Subjects with mild renal insufficiency (CKD stage 2, GFR: 60-89 mL/min)
  Interventions: Drug: PB119
- Group B (Experimental): Subjects with moderate renal insufficiency (CKD stage 3, GFR: 30-59 mL/min)
  Interventions: Drug: PB119
- Group C (Experimental): Subjects with normal renal function (GFR: ≥ 90 and < 130 mL/min)
  Interventions: Drug: PB119

INTERVENTIONS:
Drug: PB119 — Each subject received only one dose of study drug during the study period. After completing the pre-dose procedure on the morning of the first day of the study, the subjects were given a subcutaneous injection of PB-119 0.3 mL (150 μg) once in the abdomen by the study nurse. The actual time of administration will be recorded in the subject's eCRF.
  Subjects should remain on an empty stomach for at least 10 hours prior to administration.

SUMMARY:
This study is a single-dose, parallel grouping, open-label phase I clinical study to evaluate the PK characteristics and safety of single subcutaneous injection of PB-119 in subjects with different degrees of renal insufficiency and matched subjects with normal renal function.

DETAILED DESCRIPTION:
This study plans to enroll 24 subjects, which are divided into three groups: Group A: subjects with mild renal insufficiency (chronic kidney disease [CKD] stage 2); Group B: subjects with moderate renal insufficiency (CKD3 stage 3); Group C: subjects with normal renal function. The estimated glomerular filtration rate (eGFR, mL/min/1.73m2) transformed according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula should be converted into individual glomerular filtration rate (GFR, mL/min) as an indicator of CKD grading, and subjects should be stratified according to different degrees of renal function.

ELIGIBILITY:
Inclusion Criteria:

* All subjects included in this study must meet all of the following criteria:

  1. Subjects who voluntarily sign the informed consent form (ICF) before the commencement of relevant activities of this study, can understand the procedures and methods of this study, and are willing to strictly abide by the clinical study protocol to complete this study;
  2. Male subjects: Male subjects should voluntarily take effective contraceptive measures, and should not donate sperm from the screening period to 90 days after the administration of the study drug

Female subjects must meet one of the following conditions:

1. Non-fertile women
2. Fertile women should voluntarily take effective contraceptive measures from the screening period to 90 days after the administration of the study drug;
3. According to the judgment of the investigators, the subject's physical examination, vital signs examination, 12 lead ECG examination and laboratory examination indicators are suitable for participating in this study;

   Subjects in the renal insufficiency group must also meet the following criteria:
4. Male or female subjects aged between 18 and 75 years old;
5. The weight of male subjects should not be less than 50 kg and that of female subjects should not be less than 45 kg. BMI should be between 18 and 30 kg/m2 (including both end values);
6. Subjects with a diagnosis of chronic (> 3 months) and stable (no acute exacerbation due to renal function aggravated within 1 month before screening) renal injury, and a GFR measured during the screening period in line with 60 89 mL/min (mild renal insufficiency in group A) or 30-59 mL/min (moderate renal insufficiency in group B). Renal function evaluated by individual GFR converted from eGFR calculated according to the CKD-EPI formula;

   Subjects in the normal renal function group must also meet the following criteria:
7. Male or female subjects aged between 18 and 75 years old, which should be matched with age (±10 years) and gender of subjects in the renal insufficiency group;
8. The weight of male subjects should not be less than 50 kg and that of female subjects should not be less than 45 kg. BMI should be between 18 and 30 kg/m2 (including both end values), which should be matched with BMI (± 15%) of subjects in renal insufficiency group;
9. The GFR of subjects with normal renal function should be ≥ 90 and < 130 mL/min (estimated by CKD-EPI formula).

Exclusion Criteria:

* All subjects will not be included in this study if they meet any of the following criteria:

  1. Those with allergic constitution or allergic to any component in PB-119;
  2. Those with previous medical history or family history of Medullary thyroid cancer (MTC) or Multiple endocrine adenomatosis type 2 (MEN2), or serum calcitonin ≥ 50 pg/mL at screening;
  3. Those with serum amylase or lipase >3 × upper limit of normal (ULN) during the screening period or baseline period or subjects with previous diagnosis of acute/chronic pancreatitis;
  4. Those who had severe gastrointestinal diseases (such as active ulcer, gastroparesis, obstruction pyloric, inflammatory bowel disease, etc.) or underwent gastrointestinal surgery or long-term use of drugs directly affecting gastrointestinal peristalsis due to chronic gastrointestinal diseases within 6 months before screening or during the baseline period are not suitable to participate in this clinical study according to the evaluation of the investigators;
  5. Those with any type of treated or untreated malignancy (whether cured or not) within 5 years before screening or during the baseline period (except basal cell carcinoma of the skin);
  6. Those who have major diseases or surgery within 4 weeks before administration, or those who are expected to be hospitalized due to surgery or other reasons during the study period;
  7. Those with a history of drug abuse or a positive urine drug screening test within 5 years before screening;
  8. Those who smoked more than 10 cigarettes per day on average within 3 months before screening;
  9. Those with an average weekly alcohol intake of more than 14 units (female subjects) or 21 units (male subjects) (1 unit of alcohol is equivalent to 284 mL of beer, 1 glass of 125 mL of wine or 25 mL of spirits) in the 3 months prior to screening or who ingested any alcohol-containing products within 48 hours prior to administration, or those with a positive breath alcohol test;
  10. Clinical investigators who have participated in any drug or medical device within 3 months before screening (subject to administration);
  11. Those who donated blood (or lost blood) ≥ 400 mL or received blood products within 3 months before screening;
  12. Those with acute hepatitis, chronic liver disease, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × ULN and total bilirubin > 2 × ULN during the screening period or baseline period;
  13. Those who are positive for any of the hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, human immunodeficiency virus (HIV) antibody, and Treponema pallidum antibody according to the local diagnostic test;
  14. Female subjects with positive pregnancy test results during the screening period or baseline period;
  15. Those who are positive for the new coronavirus nucleic acid test during the screening period or baseline period;
  16. Those who are unable to perform venipuncture and/or tolerate catheter venous access;
  17. The investigator considers that the subject is not suitable to participate in the study due to any conditions that may cause the subject to be unable to complete the study or pose a significant risk to the subject or other factors that may reduce the possibility of enrollment;

      Subjects in the renal insufficiency group will not be included in this study if they meet any of the following criteria:
  18. Those with renal impairment with uropathy obstructive (such as urinary calculus, urinary tract obstruction caused by abdominal space-occupying lesions, etc.) or other causes unrelated to parenchymal dysfunction kidney (such as polycystic kidney, renal tumor, etc.) and/or renal diseases (such as renal artery stenosis, drugs, severe infection, insufficient blood volume, cardiac failure, etc.);
  19. Those who have received renal transplant;
  20. Those with average systolic blood pressure exceeding 80-180 mmHg (including both end values) or average diastolic blood pressure exceeding 50-100 mmHg (including both end values) or heart rate exceeding the range of 45-120 beats/min (including both end values) in the screening period or baseline period;
  21. Those who have heart failure/hypertension, respiratory, liver, gastrointestinal, endocrine (except hyperlipidemia, untreated hyperuricemia and diabetes mellitus with stable blood glucose within the past month), blood, mental/nervous and other serious diseases within 1 year before screening and are not suitable to participate in this clinical study according to the evaluation of the investigators;
  22. At screening, the therapeutic drugs and/or therapeutic drugs for other comorbidities have not been stable for at least 1 month, or there are new drugs within 1 month (except for drugs used temporarily or intermittently, such as monthly use of erythropoietin, or temporary use of diuretics, etc.), or any drugs known to change the secretion of creatinine in renal tubules within 14 days or 5 half-lives (whichever is longer) before screening, such as cimetidine, trimethoprim or sibenzoline, etc.;
  23. Subjects with diabetes mellitus who have used glucagon-like peptide-1 receptor agonist (GLP-1RA) within 1 month before administration;

      Subjects in the normal renal function group will not be included in this study if they meet any of the following criteria:
  24. Those with average systolic blood pressure exceeding 90-140 mmHg (including both end values) or average diastolic blood pressure exceeding 50-90 mmHg (including both end values) or heart rate exceeding the range of 45-120 beats/min (including both end values) in the screening period or baseline period;
  25. Subjects with fasting blood glucose (FPG) ≥ 7.0 mmol/L at screening (it can be re-tested at the judgment of the investigators);
  26. Subjects with glycosylated hemoglobin (HbA1c) ≥ 6.5% at screening;
  27. Those who have heart failure/hypertension, respiratory, liver, gastrointestinal, endocrine (except hyperlipidemia and untreated hyperuricemia), blood, mental/nervous and other serious diseases within 1 year before screening and are not suitable to participate in this clinical study according to the evaluation of the investigators;
  28. Any drug (except paracetamol/acetaminophen, including over-the-counter drugs, herbal medications and dietary supplements, such as vitamins and minerals that may affect the results of the study) have been used 14 days before administration or within 5 half-lives (whichever is longer). For subjects with hyperlipidemia, statins and/or fibrates can be used, and other lipid-regulating drugs should be evaluated by the investigators and discussed with the sponsor if necessary for exclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary PK parameters: AUC0-inf | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day13), 336 h (Day15)last detectable plasma concentration
Primary PK parameters: AUC0-t | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day13), 336 h (Day15)last detectable plasma concentration
Primary PK parameters: Cmax | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day13), 336 h (Day15)last detectable plasma concentration

SECONDARY OUTCOMES:
Secondary PK parameters: Tmax | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day13), 336 h (Day15)last detectable plasma concentration
Secondary PK parameters: T1/2 | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day3), 336 h (Day15)last detectable plasma concentration
Secondary PK parameters: Vz/F | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day3), 336 h (Day15)last detectable plasma concentration
Secondary PK parameters: CL/F | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day3), 336 h (Day15)last detectable plasma concentration
Secondary PK parameters: λz | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day3), 336 h (Day15)last detectable plasma concentration
Secondary PK parameters: MRT | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day3), 336 h (Day15)last detectable plasma concentration
Secondary PK parameters: AUC% extrapolated | Up to 336 h(Day15) post-dose
  Plasma will be collected at predose(-30 min ~ 0 min) and 2 h (Day1), 4 h (Day1), 9 h (Day1), 15 h (Day1), 24 h (Day2), 30 h (Day2), 36 h (Day2), 40 h (Day2), 48 h(Day3) ), 60 h(Day3), 72 h(Day40), 96 h(Day5), 120 h(Day6), 144 h(Day7), 192 h (Day9) , 240 h (Day11), 288 h (Day3), 336 h (Day15)last detectable plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jia Miao, MD,PhD, Principal Investigator — West China Hospital; Ping Fu, MD,PhD, Principal Investigator — West China Hospital
Locations (1):
- Jia Miao, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided